CLINICAL TRIAL: NCT05240989
Title: Correlation Between Pulmonary Rehabilitation and Thoracic Fluid Capacity: One-year Follow-up of Observation Research
Brief Title: Correlation Between Pulmonary Rehabilitation and TFC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Leader of Respiratory Therapist, Fu Jen Catholic University
Other Study IDs: PL-202008027-M
Record Dates: First submitted 2021-06-08; First posted 2022-02-15 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: COPD Received PR
Keywords: pulmonary rehabilitation; negative pressure ventilation; electrical cardiometry; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pulmonary rehabilitation — one-year regular lung rehabilitation treatment and control the intensive monitoring of hemodynamic parameters

SUMMARY:
To study the effects of lung rehabilitation on the heart's hemodynamic performance of patients with chronic bidirectional lung disease when performing routine and regular PR, and found that the effects of lung rehabilitation on the heart mechanism and patients long-term quality of life research.

DETAILED DESCRIPTION:
This study will be conducted in the Pulmonary Rehabilitation Treatment Room on the 6th floor of the Affiliated University Hospital. The acceptance conditions are: (1) treatment of chronic pulmonary obstructive pulmonary disease in the lung rehabilitation clinic, and (2) signing of the subject's consent; exclusion conditions: (1) tracheostomized patients, (2) patients who cannot perform conventional lung rehabilitation, (3) patients who use respirators at home.

The study is a prospective observational study. It is expected to include a total of 25 subjects. The study will be implemented for one year from the date of IRB adoption. Before performing PR treatment, performed the 6th and 12th Every month, routine lung function, six-minute walking tests, and non-invasive cardiac output measurements are performed. The main results are: cardiac hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* treatment of chronic pulmonary obstructive pulmonary disease in the lung rehabilitation clinic
* signing of the subject's consent

Exclusion Criteria:

* gas-cut patients
* patients who cannot perform conventional lung rehabilitation
* patients who use respirators at home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of Affiliated University Hospital
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiac hemodynamic parameters | one year
  heart rate (HR)
cardiac hemodynamic parameters | one year
  blood pressure (BP)
cardiac hemodynamic parameters | one year
  stroke volume (SV)
cardiac hemodynamic parameters | one year
  cardiac output (CO)
cardiac hemodynamic parameters | one year
  total peripheral resistance (TPR)

SECONDARY OUTCOMES:
mMRC (Modified Medical Research Council) Dyspnea Scale Dyspnea Scale | one year
  assessing the severity of breathlessness in patients with COPD
Chronic Respiratory Disease Questionnaire | one year
  The Chronic Respiratory Disease Questionnaire (CRQ) is the most commonly used disease specific measurement tool to assess health related quality of life (HRQL) in patients with chronic respiratory disease. It examines four aspects of patients' lives: dyspnoea, fatigue, emotional function, and mastery (the feeling of control over the disease and its effects).
COPD Assessment Test | one year
  measure the impact of COPD on a person's life, and how this changes over time. Patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dysnea, chest tighteness) on health status. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farias CC, Resqueti V, Dias FA, Borghi-Silva A, Arena R, Fregonezi GA. Costs and benefits of pulmonary rehabilitation in chronic obstructive pulmonary disease: a randomized controlled trial. Braz J Phys Ther. 2014 Mar-Apr;18(2):165-73. doi: 10.1590/s1413-35552012005000151. Epub 2014 May 2. PMID 24838809
- [Background] Peng DM, Zampi JD, Smith SM, Yu S, Rottach N, Lowery R, Lim HM, Riegger LQ, Schumacher KR, Rocchini A. Acute Hemodynamic Effects of Negative Extrathoracic Pressure in Fontan Physiology. Pediatr Cardiol. 2019 Dec;40(8):1633-1637. doi: 10.1007/s00246-019-02197-x. Epub 2019 Aug 29. PMID 31468061
- [Background] Huang HY, Chou PC, Joa WC, Chen LF, Sheng TF, Lin HC, Yang LY, Pan YB, Chung FT, Wang CH, Kuo HP. Pulmonary rehabilitation coupled with negative pressure ventilation decreases decline in lung function, hospitalizations, and medical cost in COPD: A 5-year study. Medicine (Baltimore). 2016 Oct;95(41):e5119. doi: 10.1097/MD.0000000000005119. PMID 27741132